CLINICAL TRIAL: NCT04166994
Title: Improving Healthcare Outcomes in American Indian and Hispanic Transplant Recipients Using Culturally-Tailored Novel Technology (IMPACT)
Brief Title: Pilot of IMPACT Intervention at the University of New Mexico
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Larissa Myaskovsky, PhD, Associate Professor, Director: CHEK-D, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-413 IMPACT
Record Dates: First submitted 2019-10-30; First posted 2019-11-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Kidney Replacement
Keywords: Diet; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACT Intervention (Experimental): Incorporate a rehabilitation approach to slowly increasing KT recipients' physical activity in addition to individualized dietary intervention at every post-transplant appointment through six months post-transplant, with follow-up at 12 months post-transplant.
  Interventions: Behavioral: Exercise and diet
- Usual Care (Other): No exercise or diet specialization.
  Interventions: Other: No Intervention: Usual Care

INTERVENTIONS:
Behavioral: Exercise and diet — IMPACT Intervention
  Arms: IMPACT Intervention
Other: No Intervention: Usual Care — No exercise or diet specialization.
  Arms: Usual Care

SUMMARY:
Kidney transplant recipients (KTR) are at greater risk of weight gain, diabetes and cardiovascular events post-transplant; but medications are limited in their effectiveness, and patients may face contraindications and unwanted side effects, given their complex post-transplant immunosuppression regimen. The investigators will pilot a randomized-controlled trial to test the feasibility and acceptability of a culturally-appropriate, multi-behavior (diet and exercise) lifestyle intervention for 20 American Indian, Hispanic/Latino(a), and White KTRs. Critical components of the pilot trial include: (a) an individually tailored exercise and diet plan with a physical therapist/exercise physiologist and a registered dietitian nutritionist, who will work closely with the post-transplant team to carefully monitor patient stability; and, (b) the use of the Twistle Patient Engagement Platform to follow-up with participants between their scheduled appointments and to collect all questionnaire data.

DETAILED DESCRIPTION:
In Improving Healthcare Outcomes in American Indian and Hispanic Transplant Recipients Using Culturally-Tailored Novel Technology (IMPACT), the investigators will pilot the feasibility and acceptability of a culturally-tailored, multi-behavior lifestyle intervention using a novel technology for 14-20 AI, HL, and White KT recipients. Because of KT recipients' varied stability immediately post-transplant, and the need to individually monitor their post-transplant immunosuppression regimen, a critical component of IMPACT will be an individually-tailored exercise and diet plan with a physical therapist/exercise physiologist and a registered dietitian nutritionist, who will work closely with the post-transplant team to carefully monitor patient stability. IMPACT will combine a personalized assessment of the patient's food preferences and access to exercise resources within their environment (based on a standard list of factors developed by the nutrition and rehabilitation experts) along with clinical specifications from the transplant team. The study is innovative because it addresses previous limitations, while adapting the intervention to meet the needs of the culturally-diverse ESKD population. The final innovation of the IMPACT Pilot is the use of the Twistle Patient Engagement Platform to follow-up with participants between their scheduled appointments, ensure adherence to the intervention, collect all questionnaire data, and enhance participant retention.

ELIGIBILITY:
Inclusion Criteria:

1. Received kidney transplant at UNMH
2. Greater than 18 years of age
3. Mentally competent

Exclusion Criteria:

1. Children under the age of 18
2. Incarcerated patients
3. Pregnant women
4. Active systemic infection
5. Non-skin malignancy or melanoma in the past 2 years
6. Known cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: Satisfaction | 12 months
  Client Satisfaction Questionnaire, rated 1-4, where higher satisfaction will indicate greater intervention acceptability
Intervention Acceptability: Usability | 12 months
  System Usability Scale, rated 1-5, where higher scores indicate ease of usability
Intervention feasibility: Retention | Through study completion, an average of 1 year
  Retention rates
Intervention feasibility: Missing data | Through study completion, an average of 1 year
  Estimates of the expected rates of missing data
Intervention feasibility: Attrition | Through study completion, an average of 1 year
  Participant attrition will be measured by counting participants who do not continue with the study
Intervention feasibility: Participation | Through study completion, an average of 1 year
  Time required for study participation during every intervention session

SECONDARY OUTCOMES:
Medical records outcomes: Weight | Through study completion, an average of 1 year
  Percent weight change
Medical records outcomes: Lipids | Through study completion, an average of 1 year
  Total cholesterol: Less than 200 mg/dL, LDL: Less than 100 mg/dL, HDL: 60 mg/dL or higher, Triglycerides: less than 150 mg/dL
Medical records outcomes: HbA1c | Through study completion, an average of 1 year
  HbA1c
Patient reported outcomes: Sleep | Baseline, 1 year
  Pittsburgh Sleep Quality Index will measure different aspects of sleep and becomes one composite score, where lower scores denote a healthier sleep quality
Patient reported outcomes: QOL | Baseline, 1 year
  We will use the PROMIS Scale v1.2 Global Health measure to assess quality of life (QOL), which includes items relevant to patients with kidney disease, including overall health, physical limitations, work, pain, energy, and emotional problems.
Patient reported outcomes: Occupational | Baseline, 1 year
  Occupational Functioning Subscale: CHART-SF rated 0-100, where higher scores indicate greater levels of participation

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Myaskovsky, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04166994/Prot_SAP_004.pdf
  • Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04166994/ICF_003.pdf